CLINICAL TRIAL: NCT01529073
Title: Phase II Clinical Trial to Evaluate the Antiviral Activity of Pegylated Interferon Plus Ribavirin Plus Nitazoxanide in Individuals With Chronic Hepatitis Due to HCV Genotype 4 and Coinfected by HIV
Brief Title: Efficacy of Pegylated Interferon Plus Ribavirin Plus Nitazoxanide in HCV Genotype 4 and HIV Coinfection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Juan Macías (Other Government)
Collaborators: Spanish National Health System (Other)
Responsible Party: Sponsor-Investigator, Juan Macías, MD, PhD, Andaluz Health Service
Organization: Andaluz Health Service (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTZSPA001; 2010-024336-42 (EudraCT Number)
Record Dates: First submitted 2012-02-05; First posted 2012-02-08 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: HCV Coinfection; HIV Infection
Keywords: HIV; genotype 4 HCV; pegylated interferon; ribavirin; nitazoxanide
MeSH Terms: conditions — HIV Infections | interventions — nitazoxanide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nitazoxanide (Experimental)
  Interventions: Drug: Nitazoxanide

INTERVENTIONS:
Drug: Nitazoxanide — Nitazoxanide 500 mg bid po for 4 weeks, followed by nitazoxanide 500 mg bid plus pegylated interferon alpha 2b 1.5 mg/kg/week sc plus weight-adjusted ribavirin po for 48 weeks.
  Other Names: Alinia; Annita; Daxon; Dexidex; Kidonax; Mitafar; Pacovanton; Paramix; Nitax; Zox; Nitazox; Niazid; Toza

SUMMARY:
Objectives: 1. Primary objective: To Evaluate the rate of sustained virological response (SVR) of pegylated interferon alfa-2b (Peg-IFN) plus ribavirin (RBV) plus nitazoxanide (NTZ) in patients coinfected by HIV and HCV genotype 4 (HCV-4), never treated before (naïve) and with a treatment failure to a standard therapy with Peg-IFN plus RBV (experienced), and to compare it with the rate of SVR of these patients with Peg-IFN plus RBV is a historical cohort. 2. Secondary objectives: In naive, as well as in experienced patients: a) To evaluate the virological activity at weeks 4 and 12 after starting the combination of Peg-IFN plus RBV plus NTZ in HIV/HCV-4-coinfected patients. b) To analyze the safety of Peg-IFN plus RBV plus NTZ in HIV/HCV-4-coinfected patients.

Design: Pilot clinical trial without control to evaluate efficacy and safety (phase II).

Patients: Individuals with HIV infection and with confirmed chronic HCV infection.

Treatment: NTZ 500 mg every 12 hours during 4 weeks, followed by NTZ 500 mg every 12 hours plus Peg-IFN plus weigh-adjusted RBV for 48 weeks. Total duration of therapy: 52 weeks.

Primary variable: The proportion of patients with HCV RNA ≤10 IU/ml 24 weeks after finishing the programmed length of treatment.

Secondary variables: 1. The frequency of individuals with HCV RNA ≤10 IU/ml 12 weeks after finishing the programmed length of treatment. 2. The proportion of patients with HCV RNA ≤10 IU/ml at 4 and 12 weeks after adding PegIFN plus RBV to NTZ. 3. The frequency of severe adverse events.

DETAILED DESCRIPTION:
Main Objective To evaluate the SVR rate of treatment with Peg-IFN alfa-2b plus RBV and NTZ in patients coinfected with HIV and HCV genotype 4, both never exposed to therapy against HCV or who failed a previous treatment with Peg-IFN plus RBV, and to compare with the SVR rate obtained in patients with Peg-IFN plus RBV in a historical cohort.

Secondary objectives: In naive, as well as in experienced patients:

1. To evaluate the virological activity at weeks 4 and 12 after starting the combination of Peg-IFN plus RBV plus NTZ in HIV/HCV-4-coinfected patients.
2. To analyze the safety of Peg-IFN plus RBV plus NTZ in HIV/HCV-4-coinfected patients.

Design Single arm pilot clinical trial to evaluate safety and efficacy (phase II).

Disease or disorder under study Coinfection with HIV and HCV genotype 4.

Drugs under study Nitazoxanide 500 mg every 12 hours for 4 weeks followed by nitazoxanide 500 mg every 12 hours plus pegylated interferon alfa-2b 1.5 mcg/kg/week and weight-adjusted ribavirin for 48 weeks.

Study Population and total number of subjects Patients infected with HIV-1 with chronic HCV genotype 4 who meet the selection criteria.

Number of patients included in the study: 45.

ELIGIBILITY:
Inclusion Criteria:

1. HIV infection.
2. Infection with HCV genotype 4.
3. No prior treatment with any interferon or no response to a previous treatment with Peg-IFN plus RBV. The lack of response will include both nonresponders, and those who showed relapse.
4. Stable antiretroviral therapy 24 weeks before starting the study drugs, with undetectable plasma HIV RNA during that period of time.
5. Commitment to use two non-hormonal contraception during the study and up to 24 weeks after treatment.
6. Acceptance to give written informed consent to participate in the trial.

Exclusion Criteria:

1. Antiretroviral therapy including didanosine, stavudine, zidovudine and abacavir.
2. Decompensated cirrhosis.
3. Presence of other significant liver diseases, including chronic hepatitis or acute hepatitis B, acute hepatitis hepatitis A, hemochromatosis or deficiency of alpha-1 antitrypsin.
4. Pregnancy and lactation.
5. Men planning pregnancy with their partners during the study and up to 24 weeks after treatment.
6. Active or uncontrolled depression, other psychiatric illness, or disease during the previous year which may, in the investigator's opinion, prevent participation in the study.
7. Previous suicide attempt.
8. Active thyroid disease or poorly controlled with treatment.
9. Previous autoimmune diseases such as inflammatory bowel disease, psoriasis serious, or rheumatoid arthritis, which may be exacerbated by interferon.
10. Chemotherapy or immunomodulatory 24 weeks before starting the study.
11. Serious illness, including cancer or unstable coronary disease, 24 weeks before starting the study.
12. Any chronic disease which, in the opinion of the investigator, may prevent complete the study.
13. Presence of acute or active opportunistic infections 48 weeks before starting the study.
14. Evidence of hepatocellular carcinoma or alpha-fetoprotein levels ≥ 50 ng / ml, unless an imaging technique shows no evidence of liver tumor, all obtained 24 weeks before starting the study.
15. Hemoglobinopathy or other conditions that may facilitate hemolysis.
16. Solid organ or bone marrow transplant.
17. Known hypersensitivity to any of the drugs under study.
18. Active consumption of drugs or alcohol in the opinion of the investigator would interfere with participation in the study. The use of methadone or other opiate replacement therapy is not considered an exclusion criterion.
19. Serious side effects from treatment with Peg-IFN plus RBV in patients with prior failure of such treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Sustained virological response | 24 weeks after finishing the scheduled treatment
  The proportion of patients with HCV RNA ≤10 IU/ml 24 weeks after finishing the programmed length of treatment (52 weeks).

SECONDARY OUTCOMES:
Safety of Peg-interferon plus ribavirin plus nitazoxanide | Every 4 weeks until 28 weeks of treatment, then every 8 weeks until the end of treatment (52 weeks)
  The proportion of patients with grade 3 or 4 adverse events according to the WHO classification.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Macías, MD, PhD, Principal Investigator — Infectious Diseases and Microbiology Unit. Hospital Universitario de Valme. Servicio Andaluz de Salud
Locations (1):
- H.U. Valme, Seville, Seville, Spain

REFERENCES:
- [Derived] Macias J, Lopez-Cortes LF, Tellez F, Recio E, Ojeda-Burgos G, Rios MJ, Rivero-Juarez A, Delgado M, Rivas-Jeremias, Pineda JA. Low Efficacy of Pegylated Interferon plus Ribavirin plus Nitazoxanide for HCV Genotype 4 and HIV Coinfection. PLoS One. 2015 Dec 7;10(12):e0143492. doi: 10.1371/journal.pone.0143492. eCollection 2015. PMID 26640956